CLINICAL TRIAL: NCT06294886
Title: Vaginal Fluid Collection Study for Endometrial Cancer Test Research and Development
Brief Title: Vaginal Fluid Collection for Detection of Endometrial Cancer
Status: Recruiting | Type: Observational
Sponsor: Innovis LLC (Industry)
Responsible Party: Sponsor
Other Study IDs: Innovis RD-2401
Record Dates: First submitted 2024-02-28; First posted 2024-03-06 (Actual); Last update posted 2024-03-07 (Actual); Status verified 2024-03

CONDITIONS: Endometrial Cancer
MeSH Terms: conditions — Endometrial Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Vaginal fluid samples
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Screening test to detect endometrial cancer and precancer — The device is designed to detect DNA biomarkers for cancer in cells shed from the lining of the uterus into vaginal fluid

SUMMARY:
The primary objective of this study is to obtain de-identified vaginal fluid specimens from participants with an endometrial tissue biopsy-based histopathological diagnosis of endometrial cancer (EC), endometrial hyperplasia (AEH) with atypia or endometrial intraepithelial neoplasia (EIN).

The samples will be used for the purpose of research and development of a new molecular diagnostic test for the detection of EC, AEH and EIN.

DETAILED DESCRIPTION:
For participants providing written informed consent to participate in the study, samples of vaginal fluid will be obtained by the Principal Investigator (PI) during a pelvic examination. All vaginal fluid samples will be collected ≥7 days after the endometrial biopsy and prior to initiating any therapeutic interventions including surgery, chemotherapy, radiation or hormonal therapy PIs will be provided with multiple, individually packaged Copan eNat® sterile sample collection kits including a swab and a transport tube containing a stabilizer and preservative medium as well as a pre-addressed shipping container and single-use tubes of sterile saline solution After vaginal fluid sample collection, the swab will be inserted into the tube for storage and subsequent shipping to the Sponsor's designated laboratory. The samples can be stored at ambient temperature and should be shipped to the designated laboratory within 24 hours of collection. Site(s) will provide the Sponsor with de-identified endometrial biopsy histopathology report and post-surgery histopathology report (if any) confirming the histopathological diagnosis of EC, AEH or EIN. The final diagnosis will be based on the most severe clinical histopathology (at diagnostic endometrial sampling or surgery.)

ELIGIBILITY:
Inclusion Criteria:

1. Women ≥18 years of age.
2. Women with endometrial tissue biopsy-based histopathological diagnosis of EC (any histology, including uterine carcinosarcoma), AEH or EIN.
3. Women whose planned surgical intervention (if any) includes hysterectomy, D&C, or hysteroscopic resection.
4. Participant understands the study procedures and can provide informed consent to participate in the study and authorization for release of relevant protected health information to the study Investigator.

   -

Exclusion Criteria:

1. Patient with recurrent and/or previously treated EC.
2. Receipt of preoperative neoadjuvant chemotherapy or radiotherapy for current EC diagnosis prior to study enrollment.
3. Prior hysterectomy.
4. Current known pregnancy diagnosis.
5. Prior or current biopsy and histopathology-proven cervical cancer.
6. The presence of concomitant biopsy and histopathology-proven cervical dysplasia.
7. Any prior pelvic or vaginal radiotherapy.
8. Any current or prior cancer diagnosis (except basal cell or squamous cell skin cancer, non-gyn) within the past 5 years.
9. Chemotherapy within the past 5 years.
10. Prior intervention to treat, or surgery with intent to completely remove, the target pathology for the current diagnosis during the current episode.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study will enroll women ≥18 years of age with an endometrial tissue biopsy-based histopathological diagnosis of endometrial cancer (EC), endometrial hyperplasia (AEH) with atypia, or endometrial intraepithelial neoplasia (EIN) presenting for management of their endometrial pathology.
Sampling Method: Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2024-02-19 (Actual); Primary Completion 2024-06-01 (Estimated); Study Completion 2024-06-01 (Estimated)

PRIMARY OUTCOMES:
Detection of endometrial cancer and precancer | 4 months
  To provide vaginal fluid specimens to Exact Sciences Corporation to allow for additional research and development of a screening device for the detection of endometrial cancer and endometrial hyperplasia with atypia.

CONTACTS AND LOCATIONS:
Overall Officials: Gregg S Britt, Study Director — Innovis LLC
Locations (1):
- Trials365, Shreveport, Louisiana, United States

IPD SHARING:
Plan to Share IPD: No